CLINICAL TRIAL: NCT01720966
Title: Adhesions After Open Versus Laparoscopic Resection of Colorectal Malignancies Detected During Liver Resection
Acronym: ALIVE
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RU-RTB-0004
Record Dates: First submitted 2012-10-24; First posted 2012-11-02 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Adhesions
Keywords: Adhesions; laparoscopy; laparotomy; liver resection; colorectal malignancy
MeSH Terms: conditions — Tissue Adhesions | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Laparoscopy: Patients who will undergo liver resection who have a laparoscopically performed colorectal resection in history. Assignment to cohort is on intention to treat of the primary operation.
  Interventions: Procedure: Liver resection
- Laparotomy: Patients who will undergo liver resection who have an open colorectal resection in history. Assignment to cohort is on intention to treat of the primary operation.
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Liver resection performed for metastatic disease from colorectal carcinoma

SUMMARY:
Rationale: Adhesion formation is a frequent complication after abdominal surgery. Adhesion formation might be reduced by laparoscopic surgery, however sound evidence is lacking. Colorectal surgery would be a good clinical model to investigate adhesion formation between open and laparoscopic surgery because of the adhesion formation propensity of colorectal surgery. However, a randomized controlled study to provide direct evidence is unlikely because of large numbers of patients needed for such a trial and the difficulty to check for adhesion formation at second surgery. Therefore we investigate adhesion formation after laparoscopic and open colorectal surgery for malignancy at liver surgery for metastases.

Objective: The aim of our study is to compare the incidence of adhesions after laparoscopic versus open surgery for colorectal malignancies during liver resection for colorectal metastases.

Study design: The study is designed as a prospective observational cohort study.

Study population: All consecutive, adult patients undergoing laparotomy or laparoscopy for intended liver resection or radio frequency ablation for liver metastases of a colorectal malignancy in whom inspection of the middle and lower abdomen is possible to map adhesions.

Main study parameters/endpoints:

* Primary endpoint is incidence of adhesions to the ventral abdominal wall around the site of the original incision.
* Secondary endpoints are episodes of bowel obstruction between index surgery and liver surgery; total incidence of adhesions; extent of adhesions; Zühlke classification of adhesions; performance of adhesiolysis; duration of adhesiolysis; peroperative complications: enterotomy, seromuscular injury, inadvertent organ injury during adhesiolysis; postoperative complications: delayed diagnosed perforation, SAE's.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This study is an observational study. The existence of adhesions will be assessed during laparotomy or laparoscopy for the treatment of liver metastases. The laparotomy is indicated for medical treatment and should not be enlarged solely for the assessment of adhesions nor will the operating time be influenced for this purpose.

Adhesions and peroperative complications have to be scored by the operating surgeon during or directly after surgery. The postoperative complications have to be scored during the postoperative course by the doctors on the ward. These assessments do not interfere with the treatment of the patients.

ELIGIBILITY:
Inclusion Criteria:

* laparotomy or laparoscopy for intended liver resection or radio frequency ablation for colorectal metastases
* laparoscopy or laparotomy for colorectal malignancy in history
* age ≥18 years

Exclusion Criteria:

* a history of abdominal surgery with a high risk of adhesions either before resection of the primary tumour or during the interval between resection of the primary tumour and liver resection. These high risk surgeries are:

  * Colorectal surgery
  * Ovarian surgery
  * Abdominal wall surgery
* mental incompetence

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing laparotomy or laparoscopy for intended liver resection or radio frequency ablation for colorectal metastases in the before mentioned centers will be assessed for eligibility. The planned number of patients will be recruited in approximately 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adhesion to ventral abdominal wall | peroperative (1 day)
  To compare the incidence of adhesions to the ventral abdominal wall in patients undergoing laparotomy or laparoscopy for intended liver resection for colorectal metastases after open versus laparoscopic resection of the primary tumour.

SECONDARY OUTCOMES:
Incidence of adhesions | peroperative (1 day)
  Total incidence of adhesions
Extent of adhesions | peroperative (1 day)
  Extent of adhesions
Adhesion Score | peroperative (1 day)
  Adhesion score according to Zühlke
Adhesiolysis | peroperative (1 day)
  need to perform adhesiolysis
Duration of adhesiolysis | peroperative (1 day)
  Duration of adhesiolysis in minutes
Inadvertent bowel injury | peroperative (1 day)
  Inadvertent bowel injury made during operation
Postoperative mobidity | 30 days
  Incidence of predetermined postoperative complications:
  * mortality
  * incisional wound infection
  * abdominal sepsis
  * pneumonia
  * urinary tract infection

OTHER OUTCOMES:
Small bowel obstruction in history | in history (up to 5 years preceeding second operation)
  Patient has episode of small bowel obstruction in medical history

CONTACTS AND LOCATIONS:
Overall Officials: Harry P van Goor, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (6):
- Netherlands (6):
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - Gelre Ziekenhuis, Apeldoorn
  - Ziekenhuis Gelderse Vallei, Ede
  - Maastricht University Medical Center, Maastricht
  - Daniel de hoed kliniek, Rotterdam
  - Maxima Medisch Centrum, Veldhoven

REFERENCES:
- [Background] ten Broek RP, Strik C, Issa Y, Bleichrodt RP, van Goor H. Adhesiolysis-related morbidity in abdominal surgery. Ann Surg. 2013 Jul;258(1):98-106. doi: 10.1097/SLA.0b013e31826f4969. PMID 23013804